CLINICAL TRIAL: NCT02729896
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Obinutuzumab in Combination With Atezolizumab Plus Polatuzumab Vedotin in Patients With Relapsed or Refractory Follicular Lymphoma and Rituximab in Combination With Atezolizumab Plus Polatuzumab Vedotin in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study Evaluating Safety and Efficacy of Obinutuzumab, Polatuzumab Vedotin (Pola), and Atezolizumab (Atezo) in Participants With Relapsed or Refractory Follicular Lymphoma (FL) and Rituximab, Atezo, and Pola in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29561; 2015-004845-25 (EudraCT Number)
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — atezolizumab; obinutuzumab; polatuzumab vedotin; Rituximab

ARMS (3):
- Dose-Escalation Phase (Experimental): During the induction treatment Cycle 1 (21-day cycles): participants will receive obinutuzumab on Days 1, 8, and 15 and Pola on Day 1; Cycles 2-6: participants will receive obinutuzumab on Day 1, Atezo on Day 1, and Pola on Day 1. This is followed by obinutuzumab on Day 1 of every other month starting with Month 1 for 24 months, during maintenance treatment for FL participants.
  Interventions: Drug: Atezolizumab [TECENTRIQ]; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin
- Expansion Phase (Experimental): For FL during the induction treatment Cycle 1 (21-day cycles): participants will receive obinutuzumab on Days 1, 8, and 15 and Pola at identified RP2D (decided from dose-escalation phase) on Day 1; Cycles 2-6: participants will receive obinutuzumab on Day 1 and Pola at RP2D on Day 1. This is followed by obinutuzumab on Day 1 of every other month starting with Month 1 for 24 months (during maintenance treatment for FL participants).
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Rituximab
- Safety Run-In Phase (Experimental): For DLBCL, during the induction treatment Cycles 1-6 (21-day cycles): participants will receive rituximab on Day 1 and Pola on Day 1.
  Interventions: Drug: Atezolizumab [TECENTRIQ]; Drug: Polatuzumab Vedotin; Drug: Rituximab

INTERVENTIONS:
Drug: Atezolizumab [TECENTRIQ] — Atezolizumab will be administered by intravenous (IV) infusion at a flat dose of 1200 milligram (mg) every 3 weeks (Q3W) on Day 1 of Cycles 2-6, given in 21-day cycles during induction treatment.
  NOTE: Atezolizumab treatment has been discontinued in all participants currently on study treatment.
  Arms: Dose-Escalation Phase; Safety Run-In Phase
Drug: Obinutuzumab — Obinutuzumab will be administered by IV infusion at a flat dose of 1000 mg on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-6, given in 21-day cycles during induction treatment, and on Day 1 of every other month during maintenance treatment (1 cycle=21 days; infusion rate starts at 50 mg/hour (hr) and increases every 30 min to a maximum of 400 mg/hr).
  Arms: Dose-Escalation Phase; Expansion Phase
Drug: Polatuzumab Vedotin — Polatuzumab vedotin will be administered by IV infusion. For relapsed or refractory FL either 1.4 mg/kilogram (kg) or 1.8 mg/kg (dose-escalation phase) and at RP2D (dose-expansion phase) on Day 1 of Cycles 1-6 will be given in 21-day cycles during induction treatment. For relapsed or refactory DLBCL, 1.8 mg/kg will be given during run-in phase and either 1.8 mg/kg or 1.4 mg/kg during the expansion phase (1 cycle=21 days; infusion rate starts with 90 min and decreases to 30 min).
Drug: Rituximab — Rituximab will be administered by IV infusion at 375 mg/m˄2 on Day 1 of Cycles 1-6 during induction treatment (1 cycle-21 days; infusion rate starts with 50 mg/hr and increases every 30 min to a maximum of 400 mg/hr).
  Arms: Expansion Phase; Safety Run-In Phase

SUMMARY:
This study will evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of obinutuzumab + Atezo + Pola in participants with relapsed or refractory (RR) FL and rituximab + Atezo + Pola in participants with RR DLBCL. The study will include an initial dose-escalation phase designed to determine the recommended Phase 2 dose (RP2D) for Pola in this treatment combination, followed by an expansion phase in which Pola will be given at the RP2D. All participants will receive induction treatment with obinutuzumab + Atezo + Pola for 6 cycles. RR FL participants achieving a complete response (CR), partial response (PR), or stable disease (SD) at the end of induction (EOI) will receive maintenance treatment with obinutuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* For obinutuzumab + Atezo + Pola treatment group: relapsed or refractory FL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-Cluster of Differentiation (CD)20 monoclonal antibody and for which no other more appropriate treatment option exists as determined by the investigator
* For rituximab + Atezo + Pola treatment group: relapsed or refractory DLBCL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody, in participants who are not eligible for second line combination (immuno-) chemotherapy and autologous stem-cell transplantation or who have failed second line combination (immuno-) chemotherapy or experienced disease progression following autologous stem-cell transplantation
* Histologically documented CD20-positive lymphoma and fluorodeoxyglucose (FDG)-avid lymphoma (that is PET-positive lymphoma) with at least one bi-dimensionally measurable lesion
* Availability of a representative tumor specimen and the corresponding pathology report for retrospective central confirmation of the diagnosis of FL or DLBCL
* For women who are not postmenopausal or surgically sterile: agreement to remain abstinent or to use contraceptive methods that result in a failure rate of less than (<) 1% per year during the treatment period for greater than or equal to (>=) 5 months after last dose of Atezo, >= 12 months after last dose of rituximab, >= 12 months after last dose of Pola, and >= 18 months after last dose of obinutuzumab
* For men: agreement to remain abstinent or to use contraceptive measures that result in a failure rate of <1% per year during the treatment period and for at least 3 months after last dose of obinutuzumab, rituximab, and Atezo and for 5 months after last dose of Pola, and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* Grade 3b follicular lymphoma
* History of transformation of indolent disease to DLBCL
* Known CD20-negative status at relapse or progression; CNS lymphoma or leptomeningeal infiltration
* Prior allogeneic stem cell transplantation (SCT), completion of autologous SCT within 100 days prior to Day 1 of Cycle 1 (D1C1)
* Prior anti-cancer therapy including: Fludarabine or alemtuzumab within 12 months prior to D1C1; radioimmunoconjugate within 12 weeks prior to D1C1; monoclonal antibody or antibody drug conjugate (ADC) within 5 half-lives or 4 weeks prior to D1C1 ; radiotherapy, chemotherapy, hormonal therapy, or targeted small-molecule therapy within 2 weeks prior to D1C1; anti-programmed death-1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4), anti-CD137/41-BB agonist, or anti-CD40 agonist antibodies
* Treatment with systemic immunosuppressive medications, including but not limited to prednisone, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to D1C1
* History of solid organ transplantation and of severe allergic or anaphylactic reaction to humanized, chimeric, or murine monoclonal antibodies
* Active infection; positive for hepatitis B surface agent (HbsAg), total hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody at screening; known history of HIV positive status, progressive multifocal leukoencephalopathy (PML), autoimmune disease
* Vaccination with a live virus vaccine or live attenuated vaccine within 28 days prior to D1C1
* Pre-existing Grade greater than (>) 1 neuropathy
* Major surgical procedure other than for diagnosis within 28 days prior to D1C1
* Inadequate hematologic function, renal function, and liver function
* Pregnant or lactating women
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (5):
  - UCLA, Los Angeles, California
  - University Miami, Miami, Florida
  - Stony Brook University Hospital, Stony Brook, New York
  - Columbia Basin Hem-Onc; Department Hematology Oncology, Kennewick, Washington
  - Robert Byrd Health Science; Dept of Medicine, Section of Hematology/Oncology, Morgantown, West Virginia
- Germany (8):
  - Städtisches Klinikum Dessau Klinik für Innere Medizin Abt. Intensivmedizin, Dessau
  - Uniklinik Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Medizinische Hochschule; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - Universitätsklinikum Jena Klinik f.Chirurgie Abt. Allgemein- und Viszeralchirurgie, Jena
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Würzburg, Würzburg
- Poland (6):
  - Szpitale Wojewodzkie w Gdyni Sp. z o.o., Gdynia
  - Wojewódzki Szpital Specjalistyczny im.MikołajaKopernika;KlinikaHematologiiUniwersytetuMedycznego, Lodz
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Medical Uni of Wroclaw; Hematology, Wroclaw

REFERENCES:
- [Derived] Topp MS, Eradat H, Florschutz A, Hochhaus A, Wrobel T, Walewski J, Knopinska-Posluszny W, Kanate AS, Lech-Maranda E, Brunnberg U, Chitra S, Nielsen TG, Sellam G, Shivhare M, Lossos IS. Anti-CD20-atezolizumab-polatuzumab vedotin in relapsed/refractory follicular and diffuse large B-cell lymphoma. J Cancer Res Clin Oncol. 2023 Feb;149(2):811-817. doi: 10.1007/s00432-021-03847-5. Epub 2022 Feb 18. PMID 35182224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 investigational centres in Germany (3), Poland (5) and USA (3).
Groups:
- Dose-Escalation FL Cohort 1.4 mg: During the induction treatment Cycle 1 (21-day cycles): participants received obinutuzumab on Days 1, 8, and 15 and pola on Day 1; Cycles 2-6: participants received 1000 milligram (mg) of obinutuzumab on Day 1, 1200 mg of atezo on Day 1, and 1.4 mg/kilogram (kg) of pola on Day 1. The 1.4 mg/kg dose was cleared by an Internal Monitoring Committee (IMC) review and escalated to 1.8 mg/kg. This was followed by obinutuzumab on Day 1 of every other month starting with Month 1 for 24 months, during maintenance treatment for FL participants.
- Dose-Escalation and Expansion FL Cohort 1.8 mg: During the induction treatment Cycle 1 (21-day cycles): participants received obinutuzumab on Days 1, 8, and 15 and pola on Day 1; Cycles 2-6: participants received 1000 mg of obinutuzumab on Day 1, 1200 mg of atezo on Day 1, and pola was escalated to 1.8 mg/kg (on Day 1); once cleared by the IMC it was declared as the recommended phase 2 dose (RP2D). This was followed by obinutuzumab on Day 1 of every other month starting with Month 1 for 24 months, during maintenance treatment for FL participants. Due to unexpected toxicity, recruitment was stopped, and atezolizumab discontinued in all treated patients. This combination will not be further developed.
- Safety Run-in and Expansion DLBCL Cohort: For DLBCL, during the induction treatment Cycles 1-6 (21-day cycles): participants received a 375 mg/m^2 IV of rituximab on Day 1 and on Day 1 of every other month during consolidation. Participants also received a 1.8 mg/kg IV of Pola on Day 1. Cycles 2-6: participants received 1200 mg of Atezo on Day 1. Due to unexpected toxicity, recruitment was stopped, and atezolizumab discontinued in all treated patients. This combination will not be further developed.
Period: Overall Study
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-in and Expansion DLBCL Cohort
Started | 3 | 10 | 23
Completed | 1 | 1 | 1
Not Completed | 2 | 9 | 22
Not completed — Death | 0 | 2 | 13
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Other | 0 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 3
Not completed — Progressive Disease | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-in and Expansion DLBCL Cohort | Total
Number analyzed (Participants) | 3 | 10 | 23 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 12 | 20
  >=65 years | 1 | 4 | 11 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (13.6) | 57.7 (11.7) | 64.3 (15.3) | 61.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 9 | 13
  Male | 3 | 6 | 14 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 3 | 9 | 18 | 30
  Unknown | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Unknown | 0 | 1 | 2 | 3
  White | 3 | 9 | 21 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CR at EOI, as Determined by the Investigator on the Basis of Positron Emission Tomography and Computed Tomography (PET-CT) Scan
Description: Tumor response assessment was performed by the investigator according to modified Lugano classification using PET/CT scan. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. 90% confidence interval (CI) for percentage of responders was calculated using Clopper-Pearson method. All PET evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 6 months)
Population: Intent-to-treat (ITT) population: All participants who enrolled in the study were included in the ITT population. Data reported for all participants for whom data were available.
Measure: Number; unit: Percentage of participants
Groups:
- Safety Run-In Phase: For DLBCL, during the induction treatment Cycles 1-6 (21-day cycles): participants received a 375 mg/m^2 IV of rituximab on Day 1 and on Day 1 of every other month during consolidation. Participants also received a 1.8 mg/kg IV of Pola on Day 1. Cycles 2-6: participants received 1200 mg of Atezo on Day 1. Due to unexpected toxicity, recruitment was stopped, and atezolizumab discontinued in all treated patients. This combination will not be further developed.
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 7 | 16
Percentage of participants | 33.33 | 14.30 | 12.50

2. Secondary Outcome: Percentage of Participants With CR at EOI, as Determined by Investigator on the Basis of CT Scans Alone
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using computed tomography (CT) scan. OR: a response of CR or PR. CR: Target nodes/nodal masses regressed to <= 1.5 cm in LDi; no extralymphatic sites of disease; organ enlargement regressed to normal; no new lesions; normal/IHC-negative bone marrow morphology. All CT evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 6 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 7 | 16
Percentage of participants | 0.00 | 57.14 | 12.50

3. Secondary Outcome: Percentage of Participants With Objective Response (CR + PR) at EOI, as Determined by the Investigator on the Basis of PET-CT Scans
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using PET/CT scan. OR: a response of CR or PR. CR: a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes & extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR with a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. All PET evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 6 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 7 | 16
Percentage of participants | 33.33 | 57.14 | 25.00

4. Secondary Outcome: Percentage of Participants With Objective Response (CR + PR) at EOI, as Determined by the Investigator on the Basis of CT Scans Alone
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using CT scan. OR: a response of CR or PR. CR: Target nodes/nodal masses regressed to <= 1.5 cm in LDi; no extralymphatic sites of disease; organ enlargement regressed to normal; no new lesions; normal/IHC-negative bone marrow morphology. PR with >= 50 percet decrease in SPD of up to six target measurable nodes and extranodal sites, a 5 mm x 5 mm default value when lesions were too small, 0 x0 mm value when lesions were no longer visible, actual measurements were used for nodes greater than 5 mm x 5 mm for lymph nodes & extralymphatic sites; absent/normal, regression for non-measured lesion; spleen enlargement regression by > 50 percent; no new lesions; reduced residual uptake in bone marrow compared to baseline. All CT evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 6 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 7 | 16
Percentage of participants | 33.33 | 57.14 | 25.00

5. Secondary Outcome: Percentage of Participants With Best Response of CR or PR During the Study, as Determined by the Investigator on the Basis of CT Scans Alone
Description: as for outcome 4
Time Frame: Baseline up to 35 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 7 | 16
Percentage of participants
  Complete response | 33.3 | 14.3 | 12.5
  Partial response | 0 | 42.9 | 12.5
  Stable disease | 33.3 | 14.3 | 6.3
  Progressive disease | 33.3 | 14.3 | 31.3
  Not available | 0 | 14.3 | 37.5

6. Secondary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the treatment. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Grading was completed according to the CTCAE, version 4.0 for severity and tumor flare reactions were graded according to NCI CTCAE v3.0.
Time Frame: Baseline up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 10 | 21
Percentage of participants | 100.00 | 100.00 | 81.00

7. Secondary Outcome: Serum Obinutuzumab Concentration
Description: pre-dose (0 hr), 30 min after EOI on Day 1 Cycle 1; pre-dose (within 5 hr), 30 min after EOI on Day 1 of Cycles 2, 4, 6; maintenance phase: pre-dose (within 5 hr) on Day 1 of Months 1, 7, 13, 19; anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 50 mg/hr and decreases every 30 min to maximum of 400 mg/hr)
Time Frame: Pre-dose (0 hr) up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg
Number analyzed (Participants) | 3 | 10
mcg/mL
  Induction cycle 1 Day 1 Pre-dose | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification. | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification.
  Induction cycle 1 Day 1 Post-dose | 308 (41.6) | 295 (171)
  Induction cycle 2 Day 1 Pre-dose | 351 (81.3) | 403 (143)
  Induction cycle 2 Day 1 Post-dose | 616 (115) | 672 (130)
  Induction cycle 4 Day 1 Pre-dose | 433 (322) | 311 (177)
  Induction cycle 4 Day 1 Post-dose: number analyzed (Participants) | 3 | 8
  Induction cycle 4 Day 1 Post-dose | 583 (189) | 619 (160)
  Induction cycle 6 Day 1 Pre-dose: number analyzed (Participants) | 3 | 9
  Induction cycle 6 Day 1 Pre-dose | 288 (123) | 308 (194)
  Induction cycle 6 Day 1 Post-dose: number analyzed (Participants) | 3 | 8
  Induction cycle 6 Day 1 Post-dose | 514 (121) | 605 (161)
  Maintenance Month 1 Day 1 Pre-dose: number analyzed (Participants) | 1 | 6
  Maintenance Month 1 Day 1 Pre-dose | 221 (NA) — Standard deviation was not estimable because there was only one sample. | 171 (131)
  Maintenance Month 7 Pre-dose: number analyzed (Participants) | 2 | 6
  Maintenance Month 7 Pre-dose | 90.4 (58.8) | 83.8 (59.6)
  Maintenance Month 13 Pre-dose: number analyzed (Participants) | 2 | 2
  Maintenance Month 13 Pre-dose | 78.8 (42.8) | 158 (1.41)
  Study drug completion or early discontinuation: number analyzed (Participants) | 0 | 1
  Study drug completion or early discontinuation |  | 37.2 (NA) — Standard deviation was not estimable because there was only one sample.
  PK and Immunogenicity follow up: number analyzed (Participants) | 2 | 3
  PK and Immunogenicity follow up | 110 (120) | 15.4 (3.20)

8. Secondary Outcome: Serum Rituximab Concentration
Description: pre-dose (0 hr), 30 min after EOI on Day 1 Cycle 1; pre-dose (within 5 hr) on Day 1 of Cycles 2, 4; pre-dose (within 5 hr), 30 min after EOI on Day 1 of Cycle 6; anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 50 mg/hr and increases every 30 min to maximum of 400 mg/hr)
Time Frame: Pre-dose (0 hr) up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Safety Run-In Phase
Number analyzed (Participants) | 21
mcg/mL
  Induction Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 9
  Induction Cycle 1 Day 1 Pre-dose | 30.4 (28.8)
  Induction Cycle 1 Day 1 Post-dose: number analyzed (Participants) | 19
  Induction Cycle 1 Day 1 Post-dose | 197 (56.9)
  Induction Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 17
  Induction Cycle 2 Day 1 Pre-dose | 43.5 (28.7)
  Induction Cycle 4 Day 1 Pre-dose: number analyzed (Participants) | 10
  Induction Cycle 4 Day 1 Pre-dose | 84.8 (35.7)
  Induction Cycle 6 Day 1 Pre-dose: number analyzed (Participants) | 13
  Induction Cycle 6 Day 1 Pre-dose | 101 (45.5)
  Induction Cycle 6 Day 1 Post-dose: number analyzed (Participants) | 12
  Induction Cycle 6 Day 1 Post-dose | 239 (42.8)

9. Secondary Outcome: Serum Atezo Concentration
Description: pre-dose (within 5 hr), 30 min after EOI on Day 1 of Cycles 2, 3, 4; pre-dose (within 5 hr) on Day 1 of Cycle 6; maintenance phase: pre-dose (within 5 hr) on Day 1 of Month 1; 30 min after EOI on Day 2 of Month 1; pre-dose (within 5 hr) on Day 1 of Month 4, 7, 13, 19; anytime during treatment discontinuation visit, 120 days after the last dose, and 1-2 years after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 60 min and decreases to 30 min)
Time Frame: Pre-dose (0 hr) up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 10 | 21
mcg/mL
  Induction Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 3 | 10 | 18
  Induction Cycle 2 Day 1 Pre-dose | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification. | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification. | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification.
  Induction Cycle 2 Day 1 Post-dose: number analyzed (Participants) | 3 | 10 | 18
  Induction Cycle 2 Day 1 Post-dose | 332 (56.7) | 365 (80.7) | 355 (78.8)
  Induction Cycle 3 Day 1 Pre-dose: number analyzed (Participants) | 3 | 9 | 14
  Induction Cycle 3 Day 1 Pre-dose | 86.9 (28.8) | 78.7 (18.4) | 79.7 (30.6)
  Induction Cycle 4 Day 1 Pre-dose: number analyzed (Participants) | 3 | 7 | 9
  Induction Cycle 4 Day 1 Pre-dose | 139 (33.1) | 125 (47.3) | 139 (56.4)
  Induction Cycle 4 Day 1 Post-dose: number analyzed (Participants) | 3 | 6 | 8
  Induction Cycle 4 Day 1 Post-dose | 462 (82.0) | 450 (136) | 489 (131)
  Induction Cycle 6 Day 1 Pre-dose: number analyzed (Participants) | 3 | 4 | 9
  Induction Cycle 6 Day 1 Pre-dose | 194 (67.7) | 181 (112) | 180 (90.6)
  Maintenance Month 1 Day 1 Pre-dose: number analyzed (Participants) | 2 | 4 | 0
  Maintenance Month 1 Day 1 Pre-dose | 100 (66.0) | 70.7 (55.5) |
  Maintenance Month 1 Day 2 Post-dose: number analyzed (Participants) | 3 | 4 | 0
  Maintenance Month 1 Day 2 Post-dose | 577 (144) | 473 (177) |
  Maintenance Month 4 Pre-dose: number analyzed (Participants) | 3 | 3 | 0
  Maintenance Month 4 Pre-dose | 240 (101) | 140 (141) |
  Maintenance Month 7 Pre-dose: number analyzed (Participants) | 2 | 2 | 0
  Maintenance Month 7 Pre-dose | 226 (134) | 221 (90.5) |
  Maintenance Month 13 Pre-dose: number analyzed (Participants) | 2 | 0 | 0
  Maintenance Month 13 Pre-dose | 106 (83.0) |  |
  Study drug completion or early discontinuation: number analyzed (Participants) | 0 | 1 | 2
  Study drug completion or early discontinuation |  | 127 (NA) — Standard deviation was not estimable because there was only one sample. | 93.0 (14.2)
  Consolidation Month 1 Day 1 Pre-dose: number analyzed (Participants) | 0 | 0 | 4
  Consolidation Month 1 Day 1 Pre-dose |  |  | 132 (43.3)
  Consolidation Month 1 Day 2 Post-dose: number analyzed (Participants) | 0 | 0 | 3
  Consolidation Month 1 Day 2 Post-dose |  |  | 503 (214)
  PK and Immunogenicity followup 120D: number analyzed (Participants) | 2 | 3 | 2
  PK and Immunogenicity followup 120D | 61.4 (60.3) | 16.8 (26.8) | 19.9 (0.778)
  PK and Immunogenicity followup 1 Year: number analyzed (Participants) | 0 | 2 | 0
  PK and Immunogenicity followup 1 Year |  | NA (NA) — The mean and standard deviation could not be calculated because they were below the limit of quantification. |

10. Secondary Outcome: Serum Pola Concentration
Description: pre-dose (0 hr) on Day 1 Cycle 1; pre-dose (within 5 hr) on Day 1 of Cycles 2, 4; maintenance phase: pre-dose (within 5 hr) on Day 1 of Months 1; anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 90 min and decreases to 30 min)
Time Frame: Pre-dose (0 hr) up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 10 | 21
mcg/mL
  Pre Day 120 Follow-up: number analyzed (Participants) | 0 | 1 | 1
  Pre Day 120 Follow-up |  | 0.136 (NA) — Standard deviation was not estimable because there was only one sample. | 2.91 (NA) — Standard deviation was not estimable because there was only one sample.
  Induction Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 0 | 1 | 1
  Induction Cycle 1 Day 1 Pre-dose |  | 0.847 (NA) — Standard deviation was not estimable because there was only one sample. | 35.9 (NA) — Standard deviation was not estimable because there was only one sample.
  Induction Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 3 | 8 | 17
  Induction Cycle 2 Day 1 Pre-dose | 2.54 (0.918) | 2.62 (1.22) | 3.37 (3.60)
  Induction Cycle 4 Day 1 Pre-dose: number analyzed (Participants) | 3 | 9 | 12
  Induction Cycle 4 Day 1 Pre-dose | 4.73 (2.10) | 4.27 (1.63) | 4.92 (2.65)
  Maintenance Month 1 Day 1 Pre-dose: number analyzed (Participants) | 2 | 3 | 0
  Maintenance Month 1 Day 1 Pre-dose | 1.30 (0.696) | 1.63 (1.75) |
  Study drug completion or early discontinuation: number analyzed (Participants) | 0 | 0 | 2
  Study drug completion or early discontinuation |  |  | 0.716 (0.200)

11. Secondary Outcome: Percentage of Participants With Human Anti-Human Antibodies (HAHAs) to Obinutuzumab
Description: Pre-dose (0 hr) on Day 1 of Cycle 1, 6, anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 50 mg/hr and increased every 30 min to maximum of 400 mg/hr)
Time Frame: Baseline up to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg
Number analyzed (Participants) | 3 | 10
Percentage of participants | 0 | 0

12. Secondary Outcome: Percentage of Participants With Human Anti-Chimeric Antibodies (HACAs) to Rituximab
Description: Pre-dose (0 hr) on Day 1 of Cycle 1, 2, 4, 6, anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 50 mg/hr and increased every 30 min to maximum of 400 mg/hr)
Time Frame: Baseline to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment. (FL cohorts not applicable as rituximab was only administered in the Safety Run- in phase).
Measure: Number; unit: Percentage of participants
Arm/Group | Safety Run-In Phase
Number analyzed (Participants) | 21
Percentage of participants
  Baseline, positive: number analyzed (Participants) | 18
  Baseline, positive | 5.6
  Baseline, negative: number analyzed (Participants) | 18
  Baseline, negative | 94.4
  Induction Cycle 2 Day 1, positive: number analyzed (Participants) | 18
  Induction Cycle 2 Day 1, positive | 5.6
  Induction Cycle 2 Day 1, negative: number analyzed (Participants) | 18
  Induction Cycle 2 Day 1, negative | 94.4
  Induction Cycle 4 Day 1: number analyzed (Participants) | 12
  Induction Cycle 4 Day 1 | 100
  Induction Cycle 6 Day 1: number analyzed (Participants) | 13
  Induction Cycle 6 Day 1 | 100
  Study drug completion: number analyzed (Participants) | 1
  Study drug completion | 100

13. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezo
Description: Pre-dose (0 hr) on Day 1 of Cycle 2, 3, 4, 6, Month 1, 4, 7, 13 and 19, anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 60 min and decreases to 30 min)
Time Frame: Baseline to 35 months
Population: The Safety Evaluable Population for this outcome measure includes participants in the DLBCL cohort who received at least one dose of any study treatment. Participants in the FL 1.4 mg and FL 1.8 mg were not anazlyed.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 10 | 21
Percentage of participants
  Induction, Cycle 2 Day 1, positive: number analyzed (Participants) | 3 | 10 | 1
  Induction, Cycle 2 Day 1, positive | 0 | 0 | 5.3
  Induction, Cycle 2 Day 1, negative: number analyzed (Participants) | 3 | 10 | 18
  Induction, Cycle 2 Day 1, negative | 0 | 0 | 94.7
  Induction, Cycle 3 Day 1, positive: number analyzed (Participants) | 3 | 10 | 1
  Induction, Cycle 3 Day 1, positive | 0 | 0 | 7.1
  Induction, Cycle 3 Day 1, negative: number analyzed (Participants) | 3 | 10 | 13
  Induction, Cycle 3 Day 1, negative | 0 | 0 | 92.9
  Induction, Cycle 4 Day 1, negative: number analyzed (Participants) | 3 | 10 | 9
  Induction, Cycle 4 Day 1, negative | 0 | 0 | 100.0
  Induction, Cycle 6 Day 1, negative: number analyzed (Participants) | 3 | 10 | 7
  Induction, Cycle 6 Day 1, negative | 0 | 0 | 100.0
  Consolidation Month 1 Day 1, negative: number analyzed (Participants) | 3 | 10 | 4
  Consolidation Month 1 Day 1, negative | 0 | 0 | 100.0
  Study drug completion, negative: number analyzed (Participants) | 3 | 10 | 2
  Study drug completion, negative | 0 | 0 | 100.0
  Atezo PK Immunogenicity Follow up (120D), negative: number analyzed (Participants) | 3 | 10 | 2
  Atezo PK Immunogenicity Follow up (120D), negative | 0 | 0 | 100.0

14. Secondary Outcome: Percentage of Participants With ATAs to Pola
Description: Pre-dose (0 hr) on Day 1 of Cycle 1, 2, 4, anytime during treatment discontinuation visit, 120 days after the last dose, and 1 year after the last dose up to 35 months (1 cycle=21 days; infusion rate: starts with 90 min and decreases to 30 min)
Time Frame: Baseline to 35 months
Population: The Safety Evaluable Population that includes patients who received at least one dose of any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-In Phase
Number analyzed (Participants) | 3 | 10 | 21
Percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization up to 35 months
Description: All adverse events that occurred on or after the first dose of study treatment are summarized by mapped term, appropriate thesaurus levels, and National Cancer Institute Common Terminology Criteria (NCI CTCAE) v4.0 grade. All-Cause Mortality is reported for the ITT population.
Arm/Group | Dose-Escalation FL Cohort 1.4 mg | Dose-Escalation and Expansion FL Cohort 1.8 mg | Safety Run-in and Expansion DLBCL Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/10 | 13/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/10 | 2/21
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation FL Cohort 1.4 mg (N=3) | Dose-Escalation and Expansion FL Cohort 1.8 mg (N=10) | Safety Run-in and Expansion DLBCL Cohort (N=21)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation FL Cohort 1.4 mg (N=3) | Dose-Escalation and Expansion FL Cohort 1.8 mg (N=10) | Safety Run-in and Expansion DLBCL Cohort (N=21)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
ANAEMIA FOLATE DEFICIENCY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 4 (7) | 3 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
SCLERITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 3 (3) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 3 (3) | 5 (5)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (3) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 4 (6) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
ORAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
RHINITIS (Infections and infestations) | 1 (4) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 2 (5) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (2) | 0 (0)
PROCALCITONIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
THYROXINE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
TRI-IODOTHYRONINE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 4 (4) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
FLUID RETENTION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
VITREOUS DEGENERATION (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT02729896/Prot_SAP_001.pdf